CLINICAL TRIAL: NCT04978545
Title: Potentializing the Effect of Calcium Hydroxide on Chemomechanical Preparation in Teeth with Post-treatment Apical Periodontitis: a Randomized Clinical Study
Brief Title: The Effect of Ca(OH)2 in Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seyda Ersahan, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Seyda Ersahan, DDS, PhD, Microbial analysis of endodontic infections in teeth with post-treatment apical periodontitis before and after medication, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-06-28; First posted 2021-07-27 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-05

CONDITIONS: Periapical Periodontitis; Polymerase Chain Reaction; Intracanal Medicament; Enterococcus Faecalis Infection
MeSH Terms: conditions — Periapical Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- calciumhydroxide (Experimental): Participants received calciumhydroxide as an intracanal medicament for a one week period
  Interventions: Other: calciumhydroxide, intracanal medicament
- chlorhexidine (Experimental): Participants received chlorhexidine gel as an intracanal medicament for a one week period
  Interventions: Other: chlorhexidine, intracanal medicament

INTERVENTIONS:
Other: calciumhydroxide, intracanal medicament — In the CH group, calcium hydroxide powder (Calxyl; OCO Products, Dirnstein, Germany) was mixed with saline in a ratio 1:1 and the paste was inserted into the canal by using lentulo spirals (Malleifer-Dentsply).
  Arms: calciumhydroxide
Other: chlorhexidine, intracanal medicament — , chlorhexidine gel 2% (Gluco-Chex 2% gel, Cerkamed, Stalowa Wola, Polland) was placed into the root canals of this group with an Ultradent Capillary Tip (Ultradent products).
  Arms: chlorhexidine

SUMMARY:
Aim of the present study was to determine the intraradicular microbiota of previously root canal-treated teeth with apical periodontitis using droplet digital polymerase chain reaction (ddPCR) and to investigate the antibacterial effectiveness of different intracanal medicaments [Ca(OH)2 and CHX] that will make classical chemomechanical preparation more effective. This superiority, parallel, randomized clinical trial was conducted in the clinic of the Endodontic Department, Faculty of Dentistry, Istanbul Medipol University, Istanbul. Sixteen patients with posttreatment apical periodontitis (one tooth each) were randomly allocated into two groups according to the intracanal medicament used (n=8, for each): calcium hydroxide (CH) and 2% chlorhexidine gel (CHX) group. Total bacterial loads, as well as the amount of Enterococcus faecalis (E.faecalis) were determined before (S1) and after (S2) chemomechanical preparation and finally, after intracanal medication (S3) by means of ddPCR.

DETAILED DESCRIPTION:
Eligibility criteria The study population consisted of 16 patients (6 women and 10 men, aged 19-63 years, mean age 34.43) presenting to the endodontic clinic at Istanbul Medipol University Dental School, for nonsurgical endodontic retreatment of teeth with apical periodontitis lesions. Sixteen previously root canal-treated teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions were included in this study. Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm. Teeth with post-treatment apical periodontitis had endodontic therapy completed more than 2 years earlier and required retreatment. Termini of the root canal fillings ranged from 0-4 mm short of the radiographic apex, with no overfilling. The teeth had intact coronal restorations, with no obvious exposure of the root-filling material to the oral cavity. Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm. Exclusion criteria were also applied, as follows: teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Root canal treatment procedures and sampling Rubber dam and an aseptic technique were used throughout the endodontic retreatment. After plaque removal and rubber dam isolation, the operative field was cleaned with 3% hydrogen peroxide and disinfected with 2.5% NaOCl solution. Then, all coronal restorations, posts and carious defects were removed and access preparation was completed when the root canal filling was properly exposed. Afterwards, the tooth (including the pulp chamber), clamp, and adjacent rubber dam were once again disinfected with 2.5% NaOCl, followed by inactivation with 10% sodium thiosulfate in order to avoid interference with bacteriological sampling. Sterility control samples (SR1) were taken from the tooth surface with a sterile Omni Swab (Whatman FTA, Sigma-Aldrich) with an ejectable head. Paper points were transferred to cryotubes containing phosphate buffered saline (PBS) solution stored at -20°C. In each case, a single root canal was sampled in order to confine the microbial evaluation to a single ecological environment. In multirooted teeth, the root with the periapical lesion was selected. If there were periapical lesions in all roots, the wider canal was selected. Two of the canals included in this study were from single-rooted teeth, 3 were buccal canals in maxillary premolars, 1 palatal canal in maxillary molar, and 10 distal canals in mandibular molars.

Old root fillings were removed using Gates-Glidden drills (Dentsply Maillefer, Ballaigues, Switzerland) and endodontic files without the use of chemical solvents. The working length (WL) was established 1 mm short of the apical foramen with an apex locator (Raypex6; VDW GmbH, Munich, Germany) and then periapical radiographs were taken to ensure that all filling material was removed. Irrigation with sterile saline solution was performed in order to remove any remaining materials and to moisten the canal prior to sample collection. Next, the canal was left filled with saline, and a small hand instrument was placed at the WL and used to gently file the canal walls. An initial microbiologic sample (S1) was taken from the root canal with sterile paper points consecutively placed at the WL. Three sterile paper points were inserted into the root canal for sampling. Each paper point was left in the canal for about 1 minute. Both the paper points and the endodontic hand instument, without the handle, were transferred to cryotubes containing 300 μL of PBS solution stored at -20°C. The samples were transferred to genetic analysis laboratory for further analysis in cold chain.

Root canals were prepared by using the Revo S files and copious irrigation with 2.5% NaOCl. The canals were apically enlarged to size 35 (AS35) at the working length. Between each instrument change, the root canal was irrigated with 5 mL of 2.5% NaOCl solution. Hence, a total of 30 mL of the irrigating solution was used. After instrumentation was completed, the smear layer was removed with 17% EDTA, which was left in the canal for 3 minutes, followed by 2.5% NaOCl. The root canal was dried with sterile paper points and flushed with 2 mL of 10% sodium thiosulfate for 1 min to inactivate the NaOCl solution. Next, a sample (S2) was taken from the canals as described for S1. After preparation, the canal was medicated with either the Ca(OH)2 or 2% chlorhexidine gel based on the study group. In the CH group, calcium hydroxide powder (Calxyl; OCO Products, Dirnstein, Germany) was mixed with saline in a ratio 1:1 and the paste was inserted into the canal by using lentulo spirals (Malleifer-Dentsply). In CHX group, chlorhexidine gel 2% (Gluco-Chex 2% gel, Cerkamed, Stalowa Wola, Polland) was placed into the root canals of this group with an Ultradent Capillary Tip (Ultradent products). All root canals of the 2 above groups were sealed with a 1-mm cotton pellet and at least 3 mm layer of temporary filling material (Cavit G; 3M ESPE AG, Seefeld, Germany).

After 7 days, the tooth was isolated, the temporary restoration removed, and disinfection procedures of the operative field were performed following the same protocol used in the first visit. A new control sample of the dental crown and dentin surrounding the pulp chamber was obtained (SR2). The medication was removed with 5 mL of saline solution and by carefully filing the canal with a master apical file. For the groups using Ca(OH)2, the calcium hydroxide antimicrobial activity was neutralized with 0.5% citric acid for a period of 1 minute, which was then removed with 5 mL of saline solution. Thus, for the groups with CHX gel, the medicament was neutralized with a mixture of 0.3% L-α-lecithin and 3% Tween 80 (Zamany A, Spangberg LS (2002) An effective method of inactivating chlorhexidine. Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology and Endodontics). Next, the root canals were irrigated with 2 mL of saline solution. The post medicament sample (S3) was obtained in the same way as the pre-medicament sample was collected and sent for the PCR analysis.

After the final sampling procedure, smear layer was removed by irrigation with 5 mL17% EDTA and then, a final rinse with 10 mL distilled water. Completion of the root canal treatment proceeded with root filling using lateral condensation of gutta-percha. Access cavities were restored with composite resin (Z250, 3M Corporation, Saint Paul, MN, USA), and a final radiograph was taken.

Total bacterial loads, as well as the amount of Enterococcus faecalis were determined before instrumentation, after instrumentation and use of the intracanal medicaments, by means of ddPCR.

Genomic DNA isolation and measurement of DNA concentration DNA was extracted using the QIAamp DNA Mini Kit (Qiagen, Germany) following the protocol recommended by the manufacturer. Before DNA isolation, samples (the tubes with paper points) were digested at 50-60°C BY vortexING for 30s in every 10 min in order to ensure disaggregation of all bacteria into the PBS solution. Afterwards, the paper points were aseptically removed from the suspension and, the bacterial suspension was pelleted by centrifugation for 10 min at 5000 g. The pellet was then resuspended in 180 µl buffer ATL supplied by QIAamp DNA Mini Kit (QIAGEN GmbH, Hilden, Germany) and 20 µl proteinase K (20 mg/ml) was added. Samples were incubated for 3 h at 56°C. Subsequently, total bacterial genomic DNA was isolated according to the protocol of the QIAamp DNA Mini Kit. The final volume of DNA solution of each sample was 150 μL and was taken into account during calculation. DNA concentration (absorbance at 260 nm) was determined with a spectrophotometer (Promega Quantifluor).

Amplification of 16S rRNA genes Primers for Universal and Enterococcus 16S rRNA genes were designed in this study. After DNA extraction of samples with QIAamp DNA Mini Kit, 700-800 bp of 16S rRNA sequences were amplified by using universal E8F forward primer (5'-AGAGTTTGATCCTGGCTCAG-3') and universal E1115R reverse primer (5'-AGGGTTGCGCTCGTTG-3') 59. The final volume of PCR reactions for each isolated bacterial strain was adjusted to 25 µl. The amplification reactions of 16S rRNA genes were performed with the following conditions. 1 cycle of predenaturation at 95°C for 3 minutes, 35 cycles of 95°C for 30 seconds, 55°C for 30 seconds, and 72°C for 30 seconds which continue with a final extension step at 72°C for 10 minutes.

The PCR products were analyzed by electrophoresis using 2% agarose gel (containing ethidium bromide) in Tris/BoratE/EDTA (TBE) buffer, with gels being analyzed under ultraviolet light (at 140V for 20 minutes). Their images were visualized under ultraviolet illumination. In addition, the control and optimization of primers to be used for ddPCR was also done in conventional PCR.

Purification and Sequencing of the 16S rRNA Gene After the PCR reactions, the purification of PCR products is done by hydrolyzing the excess primers and nucleotides with ExoSap-IT (Thermo, PN: 78201.1.ML) containing Exonuclease I and Alkaline Phosphatase enzymes. 2 µl of ExoSap-IT was mixed with 5 µl of PCR product for each sample. The ExoSap reaction is performed at 37 °C for 15 minutes (enzyme activation) followed by 15 minutes (inactivation) at 80 °C. Sequencing reactions were performed by using Bigdye™ Terminator v3.1 cycle sequencing kit (Thermo). The reactions were performed according to the kit manual for all isolated strains.

After purification of the products with Exosap, the sequence reaction was performed with BigDye Terminator v3.1 Cycle Sequencing Kit (Thermo) under the following conditions. After the sequence PCR, BigDye products were purified by colon method. Zymo ZR DNA Sequencing Clean-up Kit (Zymo Research, USA) was used for this process. All samples were purified in accordance with the protocol given in the kit and executed on the 3130XL genetic analyzer.

Droplet Digital PCR (ddPCR) Droplet Digital PCR (ddPCR) was performed using primers designed according to the 16S rRNA region specific to the total bacteria and Enterococcus faecalis species, after sequencing, absolute quantitation from the bacterial species found in the paper-point sample. Primer pairs were 16S-F-5'-AGGGAATCTTCSGCAATGGG-3' and 16S-R-5'-ACGCCCAATAAATCCGGACA-'3 for total bacteria and ENT-F-5'-CGCTTCTTTCCTCCCGAGT-3' and ENT-R-5'-GCCATGCGGCATAAACTG-3' primer pairs for Enterococcus Faecalis. In the PCR reaction, amplicons amplified with unmarked primer pairs were analyzed by labeling with Eva-Green dye. For absolute quantitation of Enterococcus and total 16S rRNA, PCR was performed with two primer pairs from the same sample. 20 µL of PCR mix containing 10 µL of 2X ddPCR EvaGreen Supermix (Bio-Rad, cat. no. 1864034), 9 µL of nuclease-free water, 0.25 µL of both forward and reverse primer and 2 ng of DNA from each sample Thermal cycling conditions were: 95◦C for 5 min, then 40 cycles of 95◦C for 30 s and 60◦C for 1 min and two final steps at 4◦C for 5 minutes and 90◦C for 5minutes with a 4◦C infinite hold. After PCR was completed, the sealed plate was transferred into the plate holder of the QX200 Droplet Reader (Bio-Rad, cat. no. 1864003).

ELIGIBILITY:
Inclusion Criteria:

* root canal-treated teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions
* Teeth with post-treatment apical periodontitis had endodontic therapy completed more than 2 years earlier and required retreatment.
* Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm.
* Termini of the root canal fillings ranged from 0-4 mm short of the radiographic apex, with no overfilling.
* The teeth had intact coronal restorations, with no obvious exposure of the root-filling material to the oral cavity.
* Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm.

Exclusion Criteria:

* teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
the sequence analysis of 16S rRNA genes by the Sanger sequencing | change from baseline to postoperative 7 days
  the Sanger sequencing
, the quantitation of total bacteria and E.faecalis in 5 different samples (SR1, S1, S2, SR2 and S3) taken from teeth were measured using the ddPCR | change from baseline to postoperative 7 days
  droplet digital PCR

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Ersahan, Assoc.Prof., Principal Investigator — IstanbulMedipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: The investigators want to share IPD including all ddPCR results with all researchers